CLINICAL TRIAL: NCT05648721
Title: The Effects of a Digital Application for Gestational Diabetes Management in Improving Patients' Compliance and Satisfaction, Glycemic Control and Pregnancy Outcomes: A Multicenter Randomized Controlled Trial
Brief Title: The Effects of a Digital Application for GDM Management in Improving Patients' Compliance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Collaborators: Bar-Ilan University, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 56-22-POR
Record Dates: First submitted 2022-11-22; First posted 2022-12-13 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2023-11

CONDITIONS: Gestational Diabetes; Pregnancy in Diabetic
Keywords: Gestational diabetes; Pregnancy; Mobile-health application; Compliance; Complications
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy in Diabetics; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile health application (Experimental): Use of GDM application for GDM management
  Interventions: Other: Datos mobile health application
- Control (Other): Regular follow-up without the GDM application
  Interventions: Other: Regular follow-up

INTERVENTIONS:
Other: Datos mobile health application — The mobile Health application will send women reminders to perform glucose tests and test results will be sent to the clinic personnel for evaluation. The clinic personnel will receive an alert if a woman does not send glucose charts or when there is an abnormality in the test results. In addition, women will be able to communicate with the clinic's personnel via chat, messages, phone calls, and video.
  Arms: Mobile health application
Other: Regular follow-up — Regular follow-up according to the local clinic protocol
  Arms: Control

SUMMARY:
Gestational diabetes mellitus (GDM) is the most prevalent complication in pregnancy. Patients' follow-up and treatment is performed in specialized GDM clinics that teach and support women in implementing lifestyle changes, blood glucose self-monitoring, and nutritional and pharmacologic therapy.

Recently, mobile health (mHealth) applications have been introduced as a resource to improve self-management and follow-up among pregnant women. The proposed study will examine the efficacy of the GDM management mHealth application in improving patients' compliance and satisfaction, glycemic control, and pregnancy outcomes.

A multicenter randomized controlled trial of women with GDM treated in the GDM clinics. Women will be randomly allocated to a research group that will use the GDM application and a control group that will receive regular follow-up without the GDM application. The primary outcome is patient compliance, defined as the actual blood glucose measurements/instructed measurements ×100. Secondary outcomes include glycemic control parameters, and maternal and neonatal complications.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women diagnosed with GDM from 13.0 gestational week
* Recruitment until 34.0 gestational week
* 18 years old and older
* Singleton pregnancy

Exclusion Criteria:

* Women with pre-gestational diabetes mellitus
* Multiple pregnancy
* Women without a Smartphone that can support the GDM application
* Refusal to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Patient compliance | During the follow up in the clinic (around 4 months)
  Defined as the actual blood glucose measurements/instructed measurements ×100

SECONDARY OUTCOMES:
Mean blood glucose of the daily glucose charts | During the follow up in the clinic (around 4 months)
Percentage of off-target glucose measurements | During the follow up in the clinic (around 4 months)
Need for pharmacotherapy for glycemic control | During the follow up in the clinic (around 4 months)
polyhydramnios | During the follow up in the clinic (around 4 months)
  At least once
Preeclampsia/gestational hypertension | During the follow up in the clinic (around 4 months)
Induction of labor | At birth
Instrumental or cesarean delivery | At birth
shoulder dystocia | At birth
Third- or fourth-degree perineal tears | At birth
Neonatal birth weight | At birth
Neonatal intensive care unit admission | A week after delivery
Hypoglycemia of the newborn | During hospitalization after delivery (around one week)
Respiratory morbidity of the newborn | During hospitalization after delivery (around one week)
Number of neonates who needed phototherapy | During hospitalization after delivery (around the first week)
Neonatal death | During hospitalization after delivery (around the first week)
Neonatal hypocalcemia | During hospitalization after delivery (around the first week)
Neonatal hypomagnesemia | During hospitalization after delivery (around the first week)
Apgar score | One and Five minutes after birth
Patients' satisfaction from the monitoring protocol | Will be evaluated up to 2 months after birth
  According to numeric rating scale (1-least satisfied, 10-most satisfied)

CONTACTS AND LOCATIONS:
Locations (5):
- Israel (5):
  - Baruch Padeh Medical center, Poriya, Tiberias, North
  - Emek medical center, Afula
  - Rambam medical center, Haifa
  - Wolfson medical center, Holon
  - Galilee medical center, Nahariya

IPD SHARING:
Plan to Share IPD: No